CLINICAL TRIAL: NCT02133846
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Sequential Cohort, Dose-Ranging Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of TPI 287 in Patients With Primary Four Repeat Tauopathies: Corticobasal Syndrome or Progressive Supranuclear Palsy
Brief Title: Safety Study of TPI-287 to Treat CBS and PSP
Acronym: TPI-287-4RT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: CBD Solutions (Unknown); Tau Consortium (Other)
Responsible Party: Principal Investigator, Adam Boxer, Adam Boxer, M.D., Ph.D., University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPI287-4RT-001
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Primary Four Repeat Tauopathies (4RT); Corticobasal Syndrome (CBS); Progressive Supranuclear Palsy (PSP); Corticobasal Degeneration (CBD)
Keywords: 4RT, CBS, PSP, CBD, TPI-287
MeSH Terms: conditions — Corticobasal Degeneration; Supranuclear Palsy, Progressive; Color Vision Defects | interventions — TPI-287

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TPI-287 low dose (Experimental): 2 mg/m2 of TPI-287 administered as a 1-hour intravenous infusion once every 3 weeks for 9 weeks (for a total of 4 infusions)
  Interventions: Drug: TPI 287 2 mg/m2; Drug: Placebo
- TPI-287 moderate dose (Experimental): 6.3 mg/m2 of TPI-287 administered as a 1-hour intravenous infusion once every 3 weeks for 9 weeks (for a total of 4 infusions).
  Interventions: Drug: Placebo; Drug: TPI-287 6.3 mg/m2
- TPI-287 high dose (Experimental): 20 mg/m2 of TPI-287 administered as a 1-hour intravenous infusion once every 3 weeks for 9 weeks (for a total of 4 infusions)
  Interventions: Drug: TPI-287 20 mg/m2; Drug: Placebo
- Placebo (Placebo Comparator): 0.9% sodium chloride as a 1-hour intravenous infusion once every 3 weeks for 9 weeks (for a total of 4 infusions)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TPI 287 2 mg/m2 — 2 mg/m2 of TPI-287 diluted with 500mL 0.9% sodium chloride. TPI-287 is a microtubule inhibitor belonging to the taxane diterpenoid (taxoid) family, and specifically to the abeotaxane class.Drug: Placebo Drug: Placebo 500mL 0.9% sodium chloride.
  Arms: TPI-287 low dose
Drug: TPI-287 20 mg/m2 — 20 mg/m2 of TPI-287 diluted with 500mL 0.9% sodium chloride. TPI-287 is a microtubule inhibitor belonging to the taxane diterpenoid (taxoid) family, and specifically to the abeotaxane class
  Arms: TPI-287 high dose
Drug: Placebo — 500mL 0.9% sodium chloride
Drug: TPI-287 6.3 mg/m2 — 6.3 mg/m2 of TPI-287 diluted with 500mL 0.9% sodium chloride. TPI-287 is a microtubule inhibitor belonging to the taxane diterpenoid (taxoid) family, and specifically to the abeotaxane class
  Arms: TPI-287 moderate dose

SUMMARY:
The purpose of this study is to determine the safety and tolerability [maximum tolerated dose (MTD) within planned dosing range] of intravenous (IV) infusions of TPI 287 administered once every 3 weeks for 9 weeks (for a total of 4 infusions) in patients with primary four repeat tauopathies (4RT), corticobasal syndrome (CBS; also called corticobasal degeneration, CBD) or progressive supranuclear palsy (PSP).

DETAILED DESCRIPTION:
The maximum tolerated dose of TPI-287 will be determined through a planned dose escalation over 3 sequential cohorts, each comprising of 11 participants randomized to either TPI-287 or placebo. TPI-287 or placebo will be administered as an intravenous infusion once every 3 weeks for 9 weeks, for a total of 4 infusions. Participants who successfully complete this phase will have the option of entering into the open label extension phase during which TPI-287 will be administered once every 3 weeks for an additional 6 weeks, for a total of 3 extra infusions.

The dose of TPI 287 will be escalated in sequential cohorts. In the low dose cohort 11 subjects each diagnosis (i.e., separate dose escalations will be performed for CBS and PSP) will be enrolled. The medium and high dose cohorts will be comprised of 11 subjects; combined CBS and PSPdiagnoses. Subjects will be assigned to cohorts in the order of study entry.

Pre-medications of diphenhyramine 25 mg (Benadryl), dexamethasone 10 mg, and famotidine 20 mg (or the H2 blocker ranitidine 50 mg) will be given IV within 60 minutes prior to each study infusion.

Safety and tolerability will be assessed through reporting of adverse events, physical and neurological testing, ECGs, as well as blood and urine analyses. Baseline and end-point measures of cognition and function, MRI brain scans, and cerebrospinal fluid (CSF) biomarker analyses will be used to determine preliminary efficacy of TPI-287 in mild-moderate AD. Pharmacokinetic and pharmacodynamic properties of TPI-287 will be calculated from blood plasma collected after the first infusion, and from CSF collected on the last visit of the placebo-controlled phase.

ELIGIBILITY:
Inclusion Criteria:

1. Between 50 and 85 years of age (inclusive);
2. Able to walk 5 steps with minimal assistance (stabilization of one arm or use of cane/walker);
3. MRI at Screening is consistent with CBS or PSP (≤ 4 microhemorrhages, and no large strokes or severe white matter disease);
4. MMSE at Screening is between 14 and 30 (inclusive);
5. FDA-approved AD medications are sometimes prescribed for CBS and PSP subjects, and are allowed as long as the dose is stable for 2 months prior to Screening. Other medications (except those listed under exclusion criteria) are allowed as long as the dose is stable for 30 days prior to Screening;
6. FDA-approved Parkinson's medications are allowed as long as the dose is stable for 2 months prior to Screening;
7. Has a reliable study partner who agrees to accompany the subject to visits, and spends at least 5 hours per week with the subject;
8. Agrees to 2 lumbar punctures;
9. Signed and dated written informed consent obtained from the subject and the subject's caregiver in accordance with local IRB regulations;
10. Males and all WCBP agree to abstain from sex or use an adequate method of contraception for the duration of the study and for 30 days after the last dose of study drug.

    Adequate contraceptive methods include those with a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as complete abstinence from sexual intercourse with a potentially fertile partner, and some double barrier methods (condom with spermicide) in conjunction with use by the partner of an intrauterine device (IUD), diaphragm with spermicide, oral contraceptives, birth control patch or vaginal ring, oral, or injectable or implanted contraceptives.

    For this study, a woman who has been surgically sterilized or who has been in a state of amenorrhea for more than two years will be deemed not to be of childbearing potential;

    For PSP Only
11. Meets National Institute of Neurological Disorders and Stroke - Society for Progressive Supranuclear Palsy (NINDS-SPSP) probable or possible PSP criteria (Litvan et al. 1996a), as modified for the Neuroprotection and Natural History in Parkinson Plus Syndromes (NNIPPS) clinical trial (Bensimon et al. 2009).

For CBS Only

11. Meets 2013 consensus criteria for possible or probable corticobasal degeneration, CBS subtype (Armstrong et al. 2013).

Exclusion Criteria:

1. Meets National Institute on Aging-Alzheimer's Association Workgroups criteria for probable AD (McKhann et al. 2011);
2. Any medical condition other than CBS or PSP that could account for cognitive deficits (e.g., active seizure disorder, stroke, vascular dementia);
3. A prominent and sustained response to levodopa therapy;
4. History of significant cardiovascular, hematologic, renal, or hepatic disease (or laboratory evidence thereof);
5. History of significant peripheral neuropathy;
6. History of major psychiatric illness or untreated depression;
7. Neutrophil count <1,500/mm3, platelets <100,000/mm3, serum creatinine >1.5 x upper limit of normal (ULN), total bilirubin >1.5 x ULN, alanine aminotransferase (ALT) >3 x ULN, aspartate aminotransferase (AST) >3 x ULN, or INR >1.2 at Screening evaluations;
8. Evidence of any clinically significant findings on Screening or baseline evaluations which, in the opinion of the Investigator would pose a safety risk or interfere with appropriate interpretation of study data;
9. Current or recent history (within four weeks prior to Screening) of a clinically significant bacterial, fungal, or mycobacterial infection;
10. Current clinically significant viral infection;
11. Major surgery within four weeks prior to Screening;
12. Unable to tolerate MRI scan at Screening;
13. Any contraindication to or unable to tolerate lumbar puncture at Screening, including use of anti-coagulant medications such as warfarin. Daily administration of 81 mg aspirin will be allowed as long as the dose is stable for 30 days prior to Screening;
14. Subjects who, in the opinion of the Investigator, are unable or unlikely to comply with the dosing schedule or study evaluations;
15. Previous exposure to microtubule inhibitors (including TPI 287) within 5 years of Screening. Treatment with microtubule inhibitors other than TPI 287 while on study will not be allowed;
16. Participation in another interventional clinical trial within 3 months of Screening;
17. Treatment with another investigational drug within 30 days of Screening. Treatment with investigational drugs other than TPI 287 while on study will not be allowed;
18. Known hypersensitivity to the inactive ingredients in the study drug;
19. Pregnant or lactating;
20. Positive pregnancy test at Screening or Baseline (Day 1);
21. Cancer within 5 years of Screening, except for non-metastatic skin cancer or non-metastatic prostate cancer not expected to cause significant morbidity or mortality within one year of baseline.

    For CBS Only:
22. History or evidence at Screening of cortical amyloid levels on 18F florbetapir PET scans consistent with underlying AD;
23. History of serum or plasma progranulin level less than one standard deviation below the normal subject mean for the laboratory performing the assay;
24. History or evidence at Screening of known disease-associated mutations in GRN or C9ORF72 genes to rule out CBS due to TDP-43 pathology;
25. History of known disease-associated mutations in ribosomal protein L3 [TDP- 43 gene (TARBP)], chromatin modifying protein 2B (CHMPB2) or valosin containing protein (VCP) genes or any other frontotemporal lobar degeneration (FTLD) causative genes discovered during the course of the trial and not associated with underlying tau pathology.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of TPI-287 in patients with primary 4RT; CBS or PSP. | 21 months (first subject enrolled to last subject completed)
  To determine the safety and tolerability [maximum tolerated dose (MTD) within planned dosing range] of intravenous (IV) infusions of TPI 287 administered once every 3 weeks for 9 weeks (for a total of 4 infusions) in patients with primary four repeat tauopathies (4RT): corticobasal syndrome (CBS) or progressive supranuclear palsy (PSP).

SECONDARY OUTCOMES:
TPI-287 levels in blood plasma and cerebrospinal fluid | 21 months (first subject enrolled to last subject completed)
  To determine the pharmacokinetic (PK) profile of TPI 287 in plasma after a single IV infusion of TPI 287 and the steady-state cerebrospinal (CSF) concentration of TPI 287 1 week after completion of the fourth infusion.

OTHER OUTCOMES:
CSF biomarkers | Screening and 1 Week after completion of the fourth study infusion
  A lumbar puncture will be performed at the screening and final visits to obtain cerebrospinal fluid (CSF). CSF biomarkers of neurodegeneration (neurofilament light chain), total tau, tau isoforms and fragments, and tau phosphopeptides.
Brain MRI scan | Screening and 2 Weeks after last double-blind infusion
  Brain MRI scans will be performed to explore effects of changes in brain network functional and structural connectivity, as well as perfusion after administration of study drug.
Degree of disability | Baseline and 1 Week after completion 4th infusion
  The Progressive Supranuclear Palsy Rating Scale (PSPRS), Schwab and England Activities of Daily Living (SEADL), clinical dementia rating scale sum of boxes (CDR-SB-FTLD) will be conducted.
Cognition | Baseline and 1 Week after 4th study infusion
  One-minute phonemic verbal fluency (PVC) test for works starting in "F", "A" and "S", Mini-Mental State Examination (MMSE)
Behavior | Screening and 2 Weeks after last infusion
  The Geriatric Depression Scale (GDS) will be conducted to determine effect a

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MD, PhD, Principal Investigator — UCSF Memory and Aging Center
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Background] Armstrong MJ, Litvan I, Lang AE, Bak TH, Bhatia KP, Borroni B, Boxer AL, Dickson DW, Grossman M, Hallett M, Josephs KA, Kertesz A, Lee SE, Miller BL, Reich SG, Riley DE, Tolosa E, Troster AI, Vidailhet M, Weiner WJ. Criteria for the diagnosis of corticobasal degeneration. Neurology. 2013 Jan 29;80(5):496-503. doi: 10.1212/WNL.0b013e31827f0fd1. PMID 23359374
- [Background] Litvan I, Agid Y, Calne D, Campbell G, Dubois B, Duvoisin RC, Goetz CG, Golbe LI, Grafman J, Growdon JH, Hallett M, Jankovic J, Quinn NP, Tolosa E, Zee DS. Clinical research criteria for the diagnosis of progressive supranuclear palsy (Steele-Richardson-Olszewski syndrome): report of the NINDS-SPSP international workshop. Neurology. 1996 Jul;47(1):1-9. doi: 10.1212/wnl.47.1.1. PMID 8710059
- [Background] Bensimon G, Ludolph A, Agid Y, Vidailhet M, Payan C, Leigh PN; NNIPPS Study Group. Riluzole treatment, survival and diagnostic criteria in Parkinson plus disorders: the NNIPPS study. Brain. 2009 Jan;132(Pt 1):156-71. doi: 10.1093/brain/awn291. Epub 2008 Nov 23. PMID 19029129
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Brunden KR, Trojanowski JQ, Smith AB 3rd, Lee VM, Ballatore C. Microtubule-stabilizing agents as potential therapeutics for neurodegenerative disease. Bioorg Med Chem. 2014 Sep 15;22(18):5040-9. doi: 10.1016/j.bmc.2013.12.046. Epub 2013 Dec 30. PMID 24433963
- [Derived] Tsai RM, Miller Z, Koestler M, Rojas JC, Ljubenkov PA, Rosen HJ, Rabinovici GD, Fagan AM, Cobigo Y, Brown JA, Jung JI, Hare E, Geldmacher DS, Natelson-Love M, McKinley EC, Luong PN, Chuu EL, Powers R, Mumford P, Wolf A, Wang P, Shamloo M, Miller BL, Roberson ED, Boxer AL. Reactions to Multiple Ascending Doses of the Microtubule Stabilizer TPI-287 in Patients With Alzheimer Disease, Progressive Supranuclear Palsy, and Corticobasal Syndrome: A Randomized Clinical Trial. JAMA Neurol. 2020 Feb 1;77(2):215-224. doi: 10.1001/jamaneurol.2019.3812. PMID 31710340